CLINICAL TRIAL: NCT03355950
Title: Comparison of Anti-sperm Antibody Levels in Inguinal Hernia Patients Who Undergo Totally Extra-peritoneal and Lichtenstein Repair
Brief Title: ASA Levels in TEP and Lichtenstein Repair Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-16-1019
Record Dates: First submitted 2017-01-30; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEP group (Active Comparator): Patients who undergo totally extraperitoneal hernia repair, TEP Repair.
  Interventions: Procedure: TEP Repair
- Lichtenstein group (Active Comparator): Patients who undergo Lichtenstein repair.
  Interventions: Procedure: Lichtenstein Repair

INTERVENTIONS:
Procedure: Lichtenstein Repair — Well defined Lichtenstein Repair for inguinal hernias
  Arms: Lichtenstein group
Procedure: TEP Repair — Laparoscopic totally extraperitoneal repair for inguianal hernias
  Arms: TEP group

SUMMARY:
The purpose of this study is to determine and compare the possible affects of two different inguinal hernia repair technique (TEP and Lichtenstein) on serum ASA levels.

DETAILED DESCRIPTION:
Antisperm antibody levels are thought to be indirect indicators of spermatic duct injuries. The investigators' ultimate goal is to draw a conclusion about the effect of the type of surgery on spermatic duct integrity. The investigators are going to collect serum samples from inguinal hernia patients before and after surgery. The investigators aim to assess the effect of surgery on antisperm antibody levels of patients who undergo Licthenstein and TEP repair. Preoperative antisperm antibody levels will serve as control levels for each patient group.

ELIGIBILITY:
Inclusion Criteria:

* to accept the terms of the randomization and all study
* to have unilateral inguinal hernia and set for an inguinal hernia repair
* to be a father

Exclusion Criteria:

* to have any kind of autoimmune disorders
* any kind of infertility history
* to have a history of inguinal and/or genital surgery and/or trauma

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Anti-sperm antibody levels after inguinal hernia surgery | Three months for each patient
  Samples will be collected before hernia surgery and three months after surgery

SECONDARY OUTCOMES:
Comparison of Anti-sperm antibody levels between inguinal hernia patients who have undergone laparoscopic totally extraperitoneal repair and Lichtenstein repair techniques | 2 years anticipated

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Coskun, MD, Prof, Study Director — Ankara Numune Research and Training Hospital
Locations (1):
- Ankara Numune Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No